CLINICAL TRIAL: NCT01975740
Title: Manual Diaphragm Release Technique Effects On Tidal Volume And Upper Rib Cage Contribution During Quiet Breathing In Elderly: A Randomized Controlled Trial
Brief Title: Manual Diaphragm Release Technique Effects On Tidal Volume in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helga Cecília Muniz de Souza, Master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Diaphragm Manual Technique
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual diaphragm release technique (Experimental)
  Interventions: Other: The manual diaphragm release technique
- Sham manual diaphragm release technique (Other)
  Interventions: Other: Sham manual diaphragm release technique

INTERVENTIONS:
Other: Sham manual diaphragm release technique
  Arms: Sham manual diaphragm release technique
Other: The manual diaphragm release technique — To perform the technique the volunteer was placed in supine position with limbs relaxed. Positioned behind the head of the volunteer, the therapist performed manual contact (pisiform, ulnar edge and the last three fingers) with the underside of the costal cartilage of the 7th, 8th, 9th and 10th rib, and guiding forearms toward the shoulders of the corresponding side. In the inspiratory phase, the therapist gently pulled the points of contact with both hands, in the direction of the head, yet slightly lateral, accompanying the elevation movement of the ribs. During exhalation, the therapist deepened contact toward the inner costal, maintaining resistance throughout the inspiratory phase. In the breaths following, the therapist sought to gain traction and smooth increase in the deepening of contacts. This maneuver was performed in two sets of ten deep breaths, with a one minute interval between them.
  Arms: Manual diaphragm release technique

SUMMARY:
Question: Does manual diaphragm release change kinematics and respiratory function of elderly subjects? Design: Randomized controlled trial with concealed allocation and double-blinding.

Participants: 17 volunteers over 60 years old randomized into two groups: 09 in the Control Group (CG) and 08 in the Intervention Group (IG).

Intervention: The manual diaphragm release technique was used on the IG, in two sets of ten deep breaths, with a one minute interval between them. The CG underwent a sham protocol (light touch), with same sets and time of interval.

Outcome measures: The groups were evaluated using spirometry, manovacuometry and optoelectronic plethysmography (OEP), in that order, before and immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* over 60 years of age;
* a body mass index (BMI) below 30 kg/m2
* non-smokers, self-declared sedentary;
* presenting a forced expiratory volume in one second (FEV1) and forced vital capacity (FVC) greater than or equal to 80% of predicted;
* the ratio between these variables (FEV1/FVC) greater than 70% in spirometry

Exclusion Criteria:

* Showed the inability to understand verbal commands in the evaluation.

Ages: 60 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Compartmental chest wall distribution | before first session
  The analysis of the regional distribution of respiratory volumes was done with Optoelectronic plethysmography (BTS Bioengineering, Italy), in which 89 reflective markers were adhered to the skin of volunteers using hypoallergenic adhesives, on particular anatomical points of the chest wall and abdomen (Aliverti and Pedotti 2003). The device emitted an infrared light on the reflective markers which was captured by eight cameras around the room, allowing the spatial determination of each marker. Thus, changes in lung volumes were calculated at each of the three compartments of the rib cage: pulmonary or upper ribcage (Rc, p), abdominal or lower ribcage (Rc, a) and abdomen (Ab). After the first OEP evaluation, a nontoxic, hypoallergenic pen was used to mark the placement of the dorsal reflective markers allowing the patient to lay in supine for the manual technique or the sham. The markers were then placed at the exact same anatomical points for reevaluation.

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressures | Before first session
  The maximal inspiratory and expiratory pressures (MIP, MEP) were obtained from the residual volume and total lung capacity, respectively, according to the criteria of the ATS/ERS (ATS/ERS, 2002) and measured using a portable digital manometer, model MVD 300 (® MDI Ltd., Brazil).
Pulmonary Function | Before first session
  To assess the participant's lung function, a portable Micro Loop 8 (Micromedical, England) spirometer was used to evaluate the forced maneuver (Miller et al 2005). The study followed the criteria of acceptability in accordance with the ATS/ERS (2005). Values of FEV1, forced vital capacity (FVC), peak expiratory flow (PEF) and FEV1/FVC were obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil